CLINICAL TRIAL: NCT04655625
Title: A Randomized, Double-blind, Placebo Controlled Phase II / III Study to Assess Safety, Immunogenicity and Efficacy of Twice Dosing of Intramuscular AG0302-COVID19 (2mg) in Healthy Adults
Brief Title: Phase II / III Study of COVID-19 DNA Vaccine (AG0302-COVID19)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AnGes, Inc. (Industry)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AG0302-COVID19-JN-02
Record Dates: First submitted 2020-11-26; First posted 2020-12-07 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: vaccine; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (AG-0302-COVID19) (Experimental)
  Interventions: Biological: Group A (AG0302-COVID19)
- Group A (Placebo) (Placebo Comparator)
  Interventions: Biological: Group A (Placebo)
- Group B (AG-0302-COVID19) (Experimental)
  Interventions: Biological: Group B (AG0302-COVID19)
- Group B (Placebo) (Placebo Comparator)
  Interventions: Biological: Group B (Placebo)

INTERVENTIONS:
Biological: Group A (AG0302-COVID19) — 2 mg of AG0302-COVID19 twice at 2-week intervals
  Arms: Group A (AG-0302-COVID19)
Biological: Group A (Placebo) — Placebo twice at 2-week intervals
  Arms: Group A (Placebo)
Biological: Group B (AG0302-COVID19) — 2 mg of AG0302-COVID19 twice at 4-week intervals
  Arms: Group B (AG-0302-COVID19)
Biological: Group B (Placebo) — Placebo twice at 4-week intervals
  Arms: Group B (Placebo)

SUMMARY:
This study will assess the safety, immunogenicity and efficacy of AG0302-COVID19 in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a Phase II /III, multi-center, randomized, double-blind, placebo controlled trial. Approximately 500 healthy volunteers, male or female, aged 18 years or older, will be randomized to one of the following two groups:

Group A: Vaccination twice at 2-week intervals (n = 250) Group B: Vaccination twice at 4-week intervals (n = 250)

Fifty subjects in each group will receive placebos.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have obtained written consent voluntarily to participate in this clinical trial
2. Subjects whose age at the time of obtaining consent is 18 years or older
3. Subjects who are negative for SARS-CoV-2 by PCR test
4. Subjects who are negative for both SARS-CoV-2 IgM antibody and SARS-CoV-2 IgG antibody by antibody test

Exclusion Criteria:

1. Subjects with symptoms of suspected COVID-19 infection (respiratory symptoms, headache, malaise, olfactory disorders, taste disorders, etc.)
2. Subjects with a history of COVID-19 (hearing from subjects)
3. Subjects who have participated in unapproved vaccine clinical trials within 1 year before the start of this study
4. Subjects with axillary temperature of 37.0 degree or higher at the time of screening and before the first vaccination
5. Subjects who have a history of anaphylaxis
6. Subjects who have a history of hypersensitivity to the ingredients of the investigational drug
7. Subjects who have a current or history of serious renal, cardiovascular, respiratory, liver, kidney, gastrointestinal, and neuropsychiatric diseases
8. Subjects with a history of convulsion or epilepsy
9. Subjects with a history of diagnosis of immunodeficiency
10. Subjects who have a close relative (within 3rd degree) of congenital immunodeficiency
11. Subjects who have current bronchial asthma
12. Subjects who have had a fever of 39.0 degrees or higher within 2 days after vaccination, or who have been suspected of having an allergy such as a systemic rash.
13. Females who wish to become pregnant from the study registration to 12 weeks after the first vaccination, and pregnant females who are breast-feeding. In addition, females who may become pregnant and their male sexual partners should use appropriate contraceptives (pill), condoms, vasectomy, tubal ligation, diaphragm, intrauterine devices, spermicides, intrauterine hormone-releasing system, etc. from the study entry date until 12 weeks after the first vaccination
14. Subjects who have participated in clinical trials of other unapproved drugs and received the investigational drug within 4 weeks before the start of this clinical trial (starting from vaccination day)
15. Subjects who have been received a live vaccine, inactivated vaccine, or toxoid within 4 weeks before the start of this clinical trial (starting from vaccination day)
16. Subjects who have been administered with drugs that affect the immune system (excluding external preparations) such as immunomodulators (DMARDs, etc.), immunosuppressants, biologics, etc. within 4 weeks before vaccination
17. Subjects who received blood transfusion or gamma globulin therapy within 12 weeks before vaccination, or high-dose gamma globulin therapy (200 mg/kg or more) within 24 weeks before vaccination
18. Subjects who have a history of overseas travel within 4 weeks before the start of the clinical trial (starting from vaccination day)
19. Subjects who are unable to comply with the clinical trial protocol and follow up (for mental, family, social or geographical reasons)
20. Subjects who are judged to be ineligible for this clinical trial by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Group A: 6 weeks Group B: 8 weeks
  Frequency and severity of each adverse event solicited local and systemic AEs from the first vaccination to 4 weeks after the second vaccination
Immunogenicity | Group A: Week 7 Group B: Week 9
  Change in Geometric mean titer (GMT) of serum anti-SARS-CoV-2 Spike (S) glycoprotein-specific antibody

SECONDARY OUTCOMES:
Change in GMT of anti-SARS-CoV-2 Spike (S) glycoprotein-specific antibody | Group A: Weeks 5, 25, 53 Group B: Weeks 7, 25, 53
Change in the neutralizing activity against pseudovirus of SARS-CoV-2 | Group A: Weeks 5, 7, 25, 53 Group B: Weeks 7, 9, 25, 53
Change in IFN-gamma production against SARS-CoV-2 spike (S) glycoprotein by T cells in peripheral blood mononuclear cells | Group A: Weeks 5, 7, 25, 53 Group B: Weeks 7, 9, 25, 53
IgG subclasses (IgG1 and IgG2) of anti-SARS-CoV-2 spike (S) glycoprotein-specific antibody | Group A: Weeks 5, 7, 25, 53 Group B: Weeks 7, 9, 25, 53
Adverse events | Group A: Week 7 through Week 53 Group B: Week 9 through Week 53
Rate of SARS-CoV-2 positive and incidence rate of COVID-19 after the first vaccination | Week 1 through Week 53

CONTACTS AND LOCATIONS:
Overall Officials: AnGes, Inc. Clinical Development, Study Director — AnGes, Inc.
Locations (8):
- Japan (8):
  - UHW Narita Hospital, Narita, Chiba
  - Medical Corporation Heishinkai OCROM Clinic, Suita, Osaka
  - Medical Corporation Tsurukamekai Shinjuku Tsurukame C linic, Shibuya-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
  - Medical Corporation Shinanokai Shinanozaka Clinic, Shinjuku-ku, Tokyo
  - Sekino Clinical Pharmacology Clinic, Toshima-ku, Tokyo
  - NISHI-UMEDA Clinic for Asian Medical Collaboration, Osaka
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No